CLINICAL TRIAL: NCT01284855
Title: A Randomized, Double-blind, Clinical Trial of Two Dose Regimens of VINS Polyvalent Antivenom (ATC J06AA03) for the Treatment of Snake Bites With Neurotoxic Envenoming in Nepal
Brief Title: Comparison of Two Dose Regimens of Snake Antivenom for the Treatment of Snake Bites Envenoming in Nepal
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CTU (Other)
Responsible Party: Sponsor-Investigator, CTU, CTU, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CER 08-192; SNF IZ70Z0 - 131 223 (Other Grant/Funding Number: Swiss National Fund)
Record Dates: First submitted 2011-01-25; First posted 2011-01-27 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Snake Bite
Keywords: neurotoxic envenoming (WHO ICD-10 T63.0)
MeSH Terms: conditions — Snake Bites | interventions — Antivenins

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low initial dose (Active Comparator): This arms corresponds to Nepal national protocol and involves the initial administration of 2 vials of antivenom over one hour followed by the slow infusion of 4 vials over 4 hours
  Interventions: Drug: Antivenom
- High initial dose (Experimental): This arms corresponds to Indian national protocol and involves the initial administration of 10 vials of antivenom over one hour followed by the slow infusion of saline over 4 hours
  Interventions: Drug: Antivenom

INTERVENTIONS:
Drug: Antivenom — Polyvalent antivenom directed against Indian spectacled cobra (N. naja), common Indian krait (B. caeruleus), saw-scaled viper (Echis carinatus) and Russell's viper.
  Other Names: VINS Bioproduct

SUMMARY:
This study aims at comparing two doses of antivenom in the treatment of snake bite envenoming. It will take place in 3 centers in rural Nepal and will involve 250 snake bite victims presenting with one or more sign of neurotoxic envenoming. The objective of the study is to generate enough scientific evidence to improve Nepal's current national guidelines for the management of snake bites.

DETAILED DESCRIPTION:
Snake bites are considered as one of the major neglected public health issues of tropical areas. They occur chiefly in developing countries and mainly affect poor rural communities. Besides the inadequate supply, distribution and accessibility of antivenom, a major problem is the absence of standardized and adequate treatment protocol. There is a significant diversity in clinical practices, in particular concerning the dose of antivenom given. Additionally, antivenom is often given even in the absence of a clear indication for envenoming. Altogether, this leads to an incredible waste of a scarce and costly resource.

In Nepal there are gross disparities in the management and outcomes of snake bite envenoming. The country's national guidelines, issued in 2004, prescribe an initial antivenom dose that is 5 times less than the one advocated by most experts. The dosage recommended by the National guidelines is not based on scientific or clinical evidence, and currently, there is confusion about the adequate dose to be administered. Some physicians follow recommendations published by experts, others follow the National guidelines, but for most, dosage is arbitrary. These discrepancies directly impact on morbidity and mortality and lead to wastage of a costly treatment that few can afford.

The principal objective of the study is to establish unequivocally which dosage regimen is the most appropriate for the treatment of snake bite neurotoxic envenoming. It is a randomized, double-blind, clinical trial comparing high and low initial doses of snake polyvalent antivenom also known as Anti Snake Venom Serum (ASVS). 250 snake bite victims showing signs of neurotoxic envenoming will be enrolled over 2 years in three health centres of Southern Nepal. Each participant will initially receive either 2 vials or 10 vials of snake polyvalent antivenom. Mortality, the proportion of patients needing assisted respiration, and the percentage of patients who show worsening of neurotoxic signs and therefore require additional doses of antivenom will be compared in both arms. The kinetics of recovery and the total consumption of antivenom will also be compared. Finally, the incidence and severity of early and late adverse reactions to antivenom will be assessed. The economical impact of snake bite envenoming will also be determined by measuring direct and indirect costs to both health services and individual victims. Because they chiefly affect agricultural workers and children, snake bites have serious economic consequences, a fact that is frequently overlooked by national authorities.

ELIGIBILITY:
Inclusion Criteria:

* History of snake bite; AND
* Age ≥ 5 years; AND
* Informed consent obtained; AND
* Showing one or more signs of neurotoxic envenoming

Exclusion Criteria:

* Subject unlikely to co-operate in the study
* Pregnant or breastfeeding women
* Patients presenting more than 24 hours after the bite
* Patients requiring ventilation support at the time of presentation
* Subjects with previous history of snake bite with envenoming
* Patients who already received antivenom before presenting to the study centre
* Patients with pre-existing neurological or muscular disorders
* Subjects with known history of allergy to horse proteins
* Patients with proven viper bites

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2011-04; Primary Completion 2012-10-15 (Actual); Study Completion 2013-03-20 (Actual)

PRIMARY OUTCOMES:
Composite endpoint: Number of patients who either 1) died, or 2) needed assisted ventilation, or 3) showed a worsening of envenoming signs during hospital stay | Participants will be followed for the duration of hospital stay, an expected average of 5 days
  The endpoint is composite and includes the number of patients who
  * die during hospitalization
  * are put under assisted ventilation during hospitalization
  * necessitate additional doses of antivenom because of a worsening of neurotoxicity.
  A worsening of neurotoxicity will be defined as the appearance of 2 new neurotoxic signs OR the appearance of a severe neurotoxic sign (i.e. loss of gag reflex or paradoxical breathing)
Number of patients with a Serious Adverse Events | Last follow-up visit (6 months after randomization)

SECONDARY OUTCOMES:
Mortality | Participants will be followed for the duration of hospital stay, an expected average of 5 days
  Number of deaths
Total amount of antivenom administered | Participants will be followed for the duration of hospital stay, an expected average of 5 days
Time to recovery | Participants will be followed for the duration of hospital stay, an expected average of 5 days
  Time between admission to the health centre and the disappearance of all neurotoxic sign s
Total cost of treatment | Last follow-up visit (6 months after randomization)
  Including direct (antivenom and other drugs costs, costs of hospitalization, and costs of Adverse Events management)and indirect costs (working days missed)
Number of patients with Adverse Events | Last follow-up visit (6 months after randomization)
Number of patients who needed assisted ventilation during hospitalization | Participants will be followed for the duration of hospital stay, an expected average of 5 days
Number of patients who showed a worsening of neurotoxicity during hospitalization | Participants will be followed for the duration of hospital stay, an expected average of 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Sanjib Sharma, MD, Principal Investigator — B. P. K. I. H. S.; François Chappuis, MD, PhD, Study Director — University Hospital, Geneva; David Warrell, MD, PhD, Study Chair — University of Oxford
Locations (3):
- Nepal (3):
  - Bharatpur Hospital, Bharatpur, Chitwan
  - Charali snake bite treatment centre, Charali, Jhapa
  - Damak red cross center, Damak, Jhapa

REFERENCES:
- [Derived] Sharma SK, Alirol E, Ghimire A, Shrestha S, Jha R, Parajuli SB, Shrestha D, Shrestha SJ, Bista A, Warrell D, Kuch U, Chappuis F, Taylor WRJ. Acute Severe Anaphylaxis in Nepali Patients with Neurotoxic Snakebite Envenoming Treated with the VINS Polyvalent Antivenom. J Trop Med. 2019 May 2;2019:2689171. doi: 10.1155/2019/2689171. eCollection 2019. PMID 31205473
- [Derived] Alirol E, Sharma SK, Ghimire A, Poncet A, Combescure C, Thapa C, Paudel VP, Adhikary K, Taylor WR, Warrell D, Kuch U, Chappuis F. Dose of antivenom for the treatment of snakebite with neurotoxic envenoming: Evidence from a randomised controlled trial in Nepal. PLoS Negl Trop Dis. 2017 May 16;11(5):e0005612. doi: 10.1371/journal.pntd.0005612. eCollection 2017 May. PMID 28510574